CLINICAL TRIAL: NCT01615146
Title: Outpatient Platelet Transfusions in Myelodysplastic Syndromes and Leukemia: The OPTIMAL Pilot
Acronym: OPTIMAL
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor recruitment
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Canadian Blood Services (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OHREB 2011500
Record Dates: First submitted 2012-06-06; First posted 2012-06-08 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2015-09

CONDITIONS: Myelodysplastic Syndrome; Leukemia
Keywords: Myelodysplasia; Leukemia; Thrombocytopenia; Platelet; transfusions; Outpatient
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia; Anemia, Refractory, with Excess of Blasts; Thrombocytopenia | interventions — Platelet Transfusion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Therapeutic Platelet Transfusion Arm (Experimental): Patients allocated to the therapeutic platelet transfusion group will not receive routine prophylactic platelet transfusions.
  Interventions: Other: Platelet Transfusion
- Prophylactic Platelet Transfusion Group (Active Comparator): Patients allocated to the prophylactic platelet transfusions will receive a platelet transfusion (a single dose of random donor platelets (4 unit pool or random donor platelets or one apheresis unit) when the measured platelet count is < 10 x 109/L.
  Interventions: Other: Platelet Transfusion

INTERVENTIONS:
Other: Platelet Transfusion — Patients allocated to the therapeutic platelet transfusion group will not receive routine prophylactic platelet transfusions. Platelet transfusions will be given to treat documented clinically relevant bleeding defined as WHO bleeding of grade 2 or greater. Patients may be transfused at the discretion of the treating physician. The indication for all platelet transfusions will be recorded by asking the ordering physician.
  Patients allocated to the prophylactic platelet transfusions will receive a platelet transfusion when the measured platelet count is < 10 x 109/L. Patients may receive additional platelet transfusions at the discretion of the treating physician. The indication for all platelet transfusions will be recorded.

SUMMARY:
As a result of the underlying disease or its therapy, it is common for patients with blood cancers to have low platelet counts. While platelet transfusions may be beneficial in preventing or treating bleeding symptoms, in circumstances where the risk of bleeding is low they may be unnecessary or even harmful. As a blood product, transfusion of platelets may be associated with infectious or allergic complications, and frequent hospital visits for transfusion may adversely affect quality of life. Additionally, the potentially overuse of platelet products places a burden on health care resources.

The benefit of the current practice of prophylactic platelet transfusions to prevent hemorrhage is unknown. The randomized data that exists is more than 25 years old and not informative given methodological limitations and the changing standards of supportive care. An alternative, therapeutic, strategy involves only administering platelets to control active bleeding.

The standard of practice in inpatients receiving high dose chemotherapy (either for acute leukemia or as part of stem cell transplantation) is prophylactic platelet transfusions. In outpatients not receiving high dose chemotherapy, the risk of bleeding is significantly lower. No randomized trials have examined the optimal platelet transfusion strategy in outpatients with blood cancers undergoing supportive or palliative therapy. Thus the potential benefit of prophylactic transfusions in the outpatient setting is unknown.

The investigators propose to perform a pilot randomized controlled trial to determine if a larger trial is possible. The ultimate goal is to determine if a strategy of therapeutic platelet transfusions is safe and effective in outpatients with blood cancers and low platelet counts.

DETAILED DESCRIPTION:
Randomization:

A local study nurse will use a web-based randomization system (permuted random blocks of two or four patients) to allocate consenting patients. Medical and research staff and investigators will be blinded to randomization scheme.

Study Duration and Follow-up:

All patients will be assigned to either a therapeutic or prophylactic platelet transfusion for a 6-month period. This period of time will allow us to assess our primary feasibility outcomes of enrollment, compliance with transfusion protocols, and completion of bleeding evaluations and quality of life questionnaires by patients.

Patients in both groups will have their CBC measured at least weekly while on study. More frequent monitoring of the platelet count may be performed at the discretion of the treating physician. The research team will clinically assess patients within 1 week (+/- 3 days) of randomization, and monthly thereafter. Patients will be asked to report any non-cutaneous grade 2 or greater bleeding immediately to their treating physicians and the study team. All the self-assessments of bleeding will be reviewed at each patient visit to ensure that all clinically relevant bleeding episodes have been captured.

Patients whose platelet count recovers to greater than 20 x 109/L for at least six weeks will be taken off the weekly platelet count monitoring as reflects clinical practice. They will continue to be monitored for the duration of the study. If their platelet count falls to 10 x 109/L or below then they will be restarted on the monitoring and previous transfusion protocol.

Data Collection:

Baseline Data - The following clinical and laboratory data will be collected at the time of enrolment: (1) demographic data, (2) diagnosis including date and disease stage, (3) prior chemotherapy, (4) ECOG performance status, (5) comorbidites, (6) previous platelet and red cell transfusions, (7) red cell transfusion history, (8) prior bleeding events, (9) quality of life (EQ5D) (10) routine bloodwork

Transfusions:

All platelet and red cell transfusions will be recorded including date and number of units. For platelet transfusions, the type of platelet product (e.g. apheresis or buffy coat) and ABO compatibility will recorded. Additionally, the indication for all transfusions (prophylactic or to treat bleeding) will be obtained from the attending physician.

Bleeding Assessment:

Participants will be asked to complete a simple bleeding questionnaire on a daily basis which has been previously tested and used in outpatients with thrombocytopenia. Patients will receive a short training session and written material on how to complete the form. A bleeding assessment will be performed at all study follow-up visits (interview, physical exam and review of daily bleeding forms). Bleeding events will be assigned a bleeding grade by the study personnel. A final bleeding grade will be assigned by an adjudication panel of 2 blinded physicians who will independently assign bleeding scores. Any discrepancies in bleeding scores will be resolved by consensus.

Quality of Life:

Quality of life will be measured using the EQ-5D. The EQ-5D is a validated tool for measurement of health-related quality of life there is a precedent for its use in transfusion medicine trials. Quality of life assessments will be performed at baseline and at all subsequent patient visits.

ELIGIBILITY:
Inclusion Criteria:

1. Adults 18 years or older with documented MDS (including MDS-subtype, CMML) or AML (as defined by WHO criteria)
2. Severe thrombocytopenia defined as a platelet count of ≤ 10 x 109/L documented on two consecutive samples at least 7 days apart.
3. Receiving outpatient-based supportive or palliative care including palliative cytoreductive, immunomodulatory or hypomethylating therapy, e.g. hydroxyurea or low dose cytarabine, lenalidomide, azacytidine, or decitabine.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 2.

Exclusion Criteria:

1. High-dose therapy in past 2 months, e.g. AML-type induction or consolidation therapy
2. Thrombocytopenia suspected to be due to immune or peripheral destruction
3. Splenomegaly, palpated at greater than 5 cm below the costal margin or greater than 20 cm on imaging
4. Alloimmune platelet refractoriness
5. Clinically relevant bleed (grade 3 or higher) within the past 3 months
6. Coagulopathy (prothrombin time or activated partial thromboplastin more than 1.5 times the upper limit of normal or fibrinogen less than 2 g/L)
7. Require anticoagulant therapy, e.g. heparin, or antiplatelet therapy, e.g. aspirin
8. Significant renal impairment (Creatinine more than 1.5 times the upper limit of normal)
9. Geographic inaccessibility resulting in the inability to comply with follow-up visits
10. Pregnant or breast-feeding
11. Unwilling or unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2012-06; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Feasibility | 18 months
  Overall enrollment, off protocol transfusions per each randomized group, total number of platelet transfusions per group and patient compliance with daily self assessment of bleeding will be evaluated.

SECONDARY OUTCOMES:
Bleeding events between therapeutic and Prophylactic transfusion groups | 6 month follow up period
  Assessments will include:
  1. Non-cutaneous Grade 2 bleeding or higher by the World Heath Organization (WHO) bleeding assessment scale 28(Appendix B)
  2. Grade 3 bleeding or higher
  3. Time from randomization to first bleeding event of grade 3 of higher
  4. Total number of red cell transfusion per group
  5. Total number of hospital days per group
  6. Number of completed daily bleeding assessments per group
  7. Quality of life
  8. Mortality

CONTACTS AND LOCATIONS:
Overall Officials: Alan Tinmouth, MD, MSc, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- the Ottawa Hospital, Ottawa, Ontario, Canada